CLINICAL TRIAL: NCT04245696
Title: Clinical Assessment of Bipolar Radiofrequency Microneedling for Improved Laxity and Lift of the Submental and Neck Tissue
Brief Title: Bipolar RF Microneedling for Improved Laxity and Lift of the Submental and Neck Tissue and Effect on Elastin
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision, no serious AEs.
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFD19002
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Skin Laxity
Keywords: RF; Micro-needling; Submental Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Group (Experimental): Single Arm: All subjects will undergo treatment for skin laxity in the submentum with a Dermal and SubQ handpiece
  Interventions: Device: Dermal Handpiece / SubQ Handpiece

INTERVENTIONS:
Device: Dermal Handpiece / SubQ Handpiece — Bipolar radiofrequency (RF) travels from the RF generator, through the electrodes and into the dermal layers beneath the surface of the skin. The microneedles of the Dermal and SubQ cartridges coupled with thermal heat will stimulate neocollagenesis and neoelastosis, aiding in the reduction of submental laxity.

SUMMARY:
This study is being conducted to evaluate the safety and efficacy of bipolar fractional radiofrequency treatment via use of the Profound System to achieve lift in lax submental (beneath the chin) and neck tissue

DETAILED DESCRIPTION:
A multi-center, blinded, non-randomized, non-controlled study

Up to 60 eligible participants will be enrolled at up to three (3) sites. Participants will receive one (1) treatment in the submental/neck area. Participants will complete follow-up visits for clinical evaluation at Day 14, 1 Month, 3 Month, and 6 Months after the study treatment. Standard photography will be obtained at Screening to the 6 Month follow-up, and 3D photography will be obtained at Screening, Month 3, and Month 6 visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults between ages 21-70 years of age.
* Desire skin laxity lift of submental and neck regions.
* Confirmed BMI ≤ 35.
* Subjects who can read, understand, and sign the Informed Consent Form.
* Subjects willing and able to comply with all study requirements.
* Fitzpatrick skin type I-VI.
* Submental fat graded by the Investigator as ≥ 1 using the Clinician-Reported Submental Fat Rating Scale (CR-SMFRS, 0=Absent (No localized submental fat evidence), 4=Extreme (Extreme submental convexity)

Exclusion Criteria:

* Active localized or systemic infections, that may alter wound healing.
* Immunocompromised subjects.
* Subjects with coagulation disorder.
* History of skin photosensitivity disorders, or use of photosensitizing drugs (e.g., tetracycline or sulfa drugs).
* Pregnant and/or lactating (All female volunteers will be advised about using birth control during the period of study).
* Excessive skin laxity on the submental and neck (Submental Skin Laxity Grade: SMSLG 4=Severe, superficial wrinkling present), or other anatomical feature for which reduction in submental fat (SMF) which may, in the judgment of the investigator, result in an aesthetically unacceptable outcome.
* Scarring in areas to be treated.
* Tattoos in the treatment areas to be treated.
* Significant open facial wounds or lesions.
* Severe or cystic acne in treatment areas.
* Current active smoker.
* Use of Accutane (Isotretinoin) within the past 6 months.
* Use of topical retinoids within 48 hours.
* Use of prescription anticoagulants.
* Pacemaker or internal defibrillator.
* History of skin disorders resulting in abnormal wound healing (i.e. keloids, extreme dry and fragile skin).
* Subjects on current oral corticosteroid therapy or within the past 6 months
* Metal implants in the treatment area.
* In the opinion of the investigator, subject is unwilling or unable to adhere to all study requirements, including application and follow-up visits.
* Subjects with a history of radiation therapy to the treatment area.
* Subject has a history of allergy to lidocaine or ester-based local anesthetics.
* Subjects with significant cardiac history or rhythm disturbance who may be unable to tolerate lidocaine with epinephrine.
* Subjects with any skin pathology or condition in the treatment area that could interfere with evaluation or with the use of typical ancillary medical treatments or care used before, during or after treatments (e.g. psoriasis, rosacea, eczema, seborrheic dermatitis, vitiligo, hyper or hypo-skin pigmentation conditions such as post inflammatory hyperpigmentation).
* Subjects who are unwilling to shave excessive hair in the treatment area that might influence or impair evaluation in the opinion of the Investigator.
* Subjects have undergone skin resurfacing or tightening treatments in the treatment area over the past year.
* Subjects have undergone dermatological treatments such as fillers and neurotoxins for the past 6 months in the treatment area.
* Subjects have undergone laser and light treatments in the treatment area over the past 3 months.
* Subjects have undergone superficial peel or microdermabrasion within 4 weeks.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Change in submental skin laxity | Baseline - Day 180 (6 months post-treatment)
  Improvement in overall lifting of treated tissue in the submental/neck region via blinded evaluation of Baseline (pre-procedure) and Day 180 (post-procedure) photographs
Occurrence, severity, and relatedness of adverse events | Baseline - Day 180 (6 months post-treatment)
  The number and level of severity of adverse events after device treatment. An assessment will also be made to determine if the adverse event is related to the study devices and/or procedure

SECONDARY OUTCOMES:
Change in submental skin laxity | Baseline - Day 90 (3 months post-treatment)
  Improvement in overall lifting of treated tissue in the submental/neck region via blinded evaluation of Baseline (pre-procedure) and Day 90 (post-procedure) photographs
Surface Area Assessment to demonstrate percentage of participants having improvement in tissue lift (> 20mm2 in submental and neck skin laxity) | Baseline vs. Day 180
  Change in submental and neck skin laxity via 3D photo-analysis
Subject assessment of improvement in skin laxity | 3 Month Follow-Up and 6 Month Follow-Up
  Improvement in skin laxity scored by subject using a 5-point Global Aesthetic Improvement Score (1=Very Much Improved, 5=Worse)
Subject satisfaction of treatment results: Subject Satisfaction scale | Day 14 - 6 Month Follow-Up
  Using a Subject Satisfaction scale, subjects will score satisfaction of treatment results (1=Not Satisfied, 5=Very Satisfied). Lower scores will show worse outcomes and higher scores will show better outcomes.
Subject assessment of pain: Numerical Pain Rating Scale | Treatment Visit
  The subjects' assessment of pain will be completed using an 11-point Numerical Pain Rating Scale (0=No pain, 10=extreme pain)

CONTACTS AND LOCATIONS:
Overall Officials: Konika Patel Schallen, MD, Principal Investigator — Candela Medical
Locations (1):
- Candela Institute of Excellence, Marlborough, Massachusetts, United States